CLINICAL TRIAL: NCT02159846
Title: The Effects of Mixed Herbs on Blood Glucose and Lipid Profile of Patients With Established Type II Diabetes Mellitus
Brief Title: Effects of Mixed Herbs on Blood Glucose and Lipid Profile in T2DM Patients
Acronym: T2DM
Status: Completed | Type: Observational
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Tahir Mahmood, Postgraduate student for the programme of, International Islamic University Malaysia
Other Study IDs: DC14-1287
Record Dates: First submitted 2014-05-22; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Herbs; Diabetes Mellitus; HbA1c; Lipid Profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test Group and Control Group: 20 patients with established T2DM were recruited from the M-OPD, HTAA, Kuantan; and equally divided into the Test and the Control groups (10 patients in each group).These patients were either fed with 4 g daily mixed herbs (on wet weight basis) or placebo (maize starch).
- Test Group & Control Group: 20 patients with established T2DM were recruited from the M-OPD, HTAA, Kuantan; and equally divided into the Test and the Control groups (10 patients in each group).These patients were either fed with 4 g daily mixed herbs (on wet weight basis) or placebo (maize starch).

SUMMARY:
The aim of this study was to evaluate the effects of mixed herbs as ad-on therapy on blood sugar and lipid profile of patients with established T2DM. A total 20 patients were consented and were equally divided into the Control and the Test groups and was fed with the Placebo or mixed herbs 4 g daily for 30 days, respectively. Blood samples were collected before and at the end of the feeding period and analyzed for the parameters namely Fasting Blood Sugar (FBS), 2 hours post prandial (2HPP) Glycosylated Hb (HbA1c) and Lipid Profile. The collected data was analyzed using SPSS Statistical Software version 12.

DETAILED DESCRIPTION:
INTRODUCTION Diabetes mellitus is a group of metabolic diseases characterized by hyperglycemia resulting from defects in insulin secretion, insulin action, or both[1]. Symptoms of marked hyperglycemia include polyuria, polydipsia, weight loss, sometimes with polyphagia, and blurred vision. Impairment of growth and susceptibility to certain infections may also accompany chronic hyperglycemia[ 2]. Several pathogenic processes are involved in the development of diabetes. These range from autoimmune destruction of the β-cells of the pancreas with consequent insulin deficiency to abnormalities that result in resistance to insulin action . Patients with diabetes have an increased incidence of atherosclerotic cardiovascular, peripheral arterial, and cerebrovascular disease. Hypertension and abnormalities of lipoprotein metabolism are often found in people with diabetes[3].

The vast majority of cases of diabetes fall into two broad etiopathogenetic categories called type 1 diabetes mellitus (T1DM) and type 2 diabetes mellitus . In T1DM, the cause is an absolute deficiency of insulin secretion. In the other, much more prevalent category, T2DM, the cause is a combination of resistance to insulin action and an inadequate compensatory insulin secretory response [4].

Despite considerable progress in the treatment of diabetes mellitus, it's prevalence is rising globally in an exponential rate to an extent that it is now the most severe pandemic of the 21st century. World Health Organization (WHO) estimated that the prevalence of diabetes for all age-groups worldwide, will increase from 2.8% in 2000 to 4.4% in 2030 whereby the total number of people with diabetes is projected to rise from 171 million in 2000, to 366 million in 2030[5].

Conventionally, insulin-dependent diabetes mellitus is treated with exogenous insulin and non insulin-dependent diabetes mellitus with synthetic oral hypoglycemic agents (OHA) like sulphonylureas and biguanides [6,7].Insulin therapy affords glycemic control in type 1 diabetes, yet its shortcomings such as ineffectiveness on oral administration, short shelf life, the requirement of constant refrigeration, fatal hypoglycemia in event of excess dosage, reluctance of patients to take insulin injection and above all, the development of resistance due to prolonged administration, limits its usage[8]. Similarly, treatment of T2DM patients with sulfonylureas and biguanides, is also associated with side effects [9].

For various reasons in recent years, the popularity of alternative medicine has increased. Surveys conducted in Australia and United States indicate that almost 48.5% and 34% of the respondents in the respective countries, had used at least one form of unconventional therapy, including herbal medicine[10].Natural materials like herbs and spices today seem to be used widely as traditional remedies for certain diseases. Spices which are added, during preparation of foods, for taste and aroma have been shown to be effective in the control of hyperglycemia both in animals and human studies[11]. Several studies conducted throughout the world, recognized the blood glucose lowering effects of herbs and spices both in animals as well as in human beings. Bunching Onion is a flavor and taste enhancer and contains many health promoting compounds that can lower, low density lipoprotein cholesterol (LDL-c) and raise high density lipoprotein cholesterol (HDL-c) level, prevent cancer, and stabilize blood sugar levels[12]. Similarly Holy Basil contains an essential oil that possesses antibacterial, antioxidant, anti-inflammatory and immune modulating effects, as well as blood sugar lowering properties in diabetic patients . Curry Leaves is an inhibitor of pancreatic enzyme α-amylase. This enzyme degrades starch to glucose in the gastrointestinal tract, which is then released to the blood stream. So by inhibiting the α-amylase enzyme, the leaves are able to prevent the degradation of starches to simple sugar (glucose), thus helping to control the hyperglycemia in patients with T2DM[13]. Onion (Allium cepa) is a common vegetable. Onion bulb and leaves are part of diet. Ether soluble fraction of onion (0.25mg/kg, orally) has been observed to lower blood sugar level in normal rabbits and exhibited potent antioxidant activity[14]. In a clinical study, treatment of diabetic patients by juice of Allium cepa bulb, controlled the blood sugar level[15]. Dipropyl-disulphideoxide and onion oil produced significant hypoglycemic effect[16]. A sulphur containing amino acid, S-methyl-cystein-sulphoxide (at a dose of 200mg/kg for 45 days) from onion showed a potent hypoglycemic activity in alloxan induced diabetic rats[17]. S-allyl-cystein-sulphoxide from onion significantly reduced blood glucose level of alloxan induced diabetic rats[18]. Prolonged administration of freeze dried onion powder (3%) with a diet produced anti-hyperglycemic, hypolipidemic and antioxidant activity in STZ diabetic rats[19]. Allium cepa juice (0.4g/100g for 4 weeks) exhibited anti-hyperglycemic and antioxidant effect in alloxan induced diabetic rats, it also repaired hepatic and renal damage caused by alloxan[20].Coriander has been used for many years to lower blood glucose in traditional herbal medicine. It has been reported that streptozotocin induced diabetic mice were fed with coriander in feed or drinking water caused a significant reduction in blood glucose[21].The anti-diabetic, hypolipidaemic and antioxidant activities of aniseeds (star anise) and coriander seeds were compared in T2DM patients. The seed powders (5 g/day) were administered to two groups of T2DM patients for 60 days. The results indicated 36% decrease in fasting blood glucose in aniseed treated, and 13%decrease in coriander treated T2DM patients, while 11% rise of fasting blood glucose in the control group. Significant decrease in serum cholesterol and triglycerides in aniseed treated and coriander seed treated patients was also observed. Both seeds have anti diabetic, hypolipidemic and antioxidant effects in diabetic patients[22].

Methodology This study was conducted at Medical Out Patient Department (M-OPD), HTAA, Kuantan, and Department of Nutrition Sciences, Kulliyyah of Allied Health Sciences, International Islamic University Malaysia (IIUM), Kuantan.

In the present study, 20 patients of T2DM were recruited from the M-OPD, HTAA, Kuantan; and equally divided into the control and the test groups. These patients were either fed with placebo (maize starch) or 4 g daily mixed herbs (on wet weight basis). Informed consent was obtained from all patients. This study was submitted to the Kulliyyah Postgraduate and Research Committee (KPGRC) for approval and subsequently to the IIUM Research Ethics Committee (IREC) and Clinical Research Committee (CRC).

The four types of herbs namely, coriander leaves (Coriandrum sativum), bunching onion (Alliumfistulosum L.), curry leaves (Murraya koenigii), and holy basil leaves (Ocimum tenuiflorum, also known as Ocimum sanctum), purchased from the local market/supplier, and thoroughly cleaned. These were then weighed and freeze-dried, weighed again and the weight loss was determined. The freeze dried herbs were ground with coffee mill and appropriate amounts were encapsulated to be offered to the patients. The consumption of the capsules was spread over the day and the numbers of capsules to be consumed per day were tailored to 4 g of wet herbs. The total duration of the trial was 30 days.

The herbs used in the trial,are not new to the patients, as each one is being used among all the communities in Malaysia for decades in preparation of their food daily, the only thing new was to observe the dose effects of these on the blood sugar and lipid profile of T2DM patients.

Data Collection All the patients were requested to provide the blood samples on Day 0, and Day 31, for the analysis of various parameters, to assess the possible effects induced by the consumption of mixed herbs.

Blood Sample Analysis The blood sample collected was immediately processed and analyzed at Biochemistry Laboratory of HTAA, for FBS, 2HPP, HbA1c, and lipid profile using appropriate kits respectively.

Statistical Analysis The current study design was Quasi-experimental study design on registered T2DM patients. Two-way ANOVA was used for statistical analysis. Furthermore, the data was expressed as mean ± SD and the difference in the means was ascertained at 95 % confidence interval (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

* The patients having established T2DM, adult, both sexes were included in the study.

Exclusion Criteria:

* The patients having T1DM, allergy or intolerant to herbs, consuming other herbal supplements and pregnant women with/without gestational diabetes mellitus (GDM) were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the present study, 20 patients with established T2DM were recruited from the M-OPD, HTAA, Kuantan; and equally divided into the control and the test groups (10 patients in each group).These patients were either fed with placebo (maize starch) or 4 g daily mixed herbs (on wet weight basis).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Allergy or hypersensitivity to preparation | within the consumption period (30 days)

CONTACTS AND LOCATIONS:
Overall Officials: TAHIR MAHMOOD, M.B;B.S, Principal Investigator — Ministry of Health
Locations (1):
- Medical Out-Patient Department (M-OPD),Hospital Tengku Ampuan Afzan Kuantan., Kuantan, Pahang, Malaysia